CLINICAL TRIAL: NCT04511923
Title: Can Nebulised HepArin Reduce acuTE Lung Injury in Patients With SARS-CoV-2 Requiring Respiratory Support in Ireland
Brief Title: Nebulised Heparin to Reduce COVID-19 Induced Acute Lung Injury
Acronym: CHARTER-Irl
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor, Anaesthesia and Intensive Care Medicine, School of Medicine, NUI Galway; Consultant, Anaesthesia and ICM, Galway University Hospitals; Vice-Dean Research, College of Medicine, Nursing, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUIG-2020-003
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Covid19; ARDS, Human; Lung Injury, Acute; Ventilation Perfusion Mismatch
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention): Standard care
- Heparin (Experimental): Standard care plus nebulised unfractionated heparin 25000 units every 6 hours for 10 days
  Interventions: Drug: Nebulised heparin

INTERVENTIONS:
Drug: Nebulised heparin — Nebulised unfractionated heparin 25000 units administered 6 hourly for 10 days
  Arms: Heparin

SUMMARY:
The investigators present a randomised open label phase Ib/IIa trial of nebulised unfractionated heparin to evaluate the effect of nebulised unfractionated heparin on the procoagulant response in ICU patients with SARS-CoV-2 requiring advanced respiratory support. As this is one of the first studies of nebulised heparin in COVID 19 lung disease the investigators will assess safety as a co-primary outcome.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, a patient must satisfy all these inclusion criteria:

1. Confirmed or suspected COVID-19. Note, if 'suspected', results must be pending or testing intended
2. Ability to obtain informed consent/assent to participate in study
3. Age 18 years or older
4. Requiring high flow nasal oxygen or positive pressure ventilator support or invasive mechanical ventilation for a time period of no greater than 48 hours
5. D-dimers > 200 ng/ml
6. PaO2 to FIO2 ratio less than or equal to 300
7. Acute opacities on chest imaging affecting at least one lung quadrant. Note 'Acute opacities' do not include effusions, lobar/lung collapse or nodules
8. Currently in a higher level of care area designated for inpatient care of patients where therapies including non-positive pressure ventilatory support can be provided.

Exclusion criteria

To be eligible, a patient must have none of these exclusion criteria:

1. Enrolled in another clinical trial that is unapproved for co-enrolment
2. Heparin allergy or heparin-induced thrombocytopaenia
3. APTT > 100 seconds
4. Platelet count < 50 x 109 per L
5. Pulmonary bleeding, which is frank bleeding in the trachea, bronchi or lungs with repeated haemoptysis or requiring repeated suctioning
6. Uncontrolled bleeding
7. Pregnant or suspected pregnancy (Urine or serum HCG will be recorded)
8. Receiving or about to commence ECMO or HFOV
9. Myopathy, spinal cord injury, or nerve injury or disease with a likely prolonged incapacity to breathe independently e.g. Guillain-Barre syndrome
10. Usually receives home oxygen
11. Dependent on others for personal care due to physical or cognitive decline (pre-morbid status)
12. Death is imminent or inevitable within 24 hours
13. The clinical team would not be able to set up the study nebuliser and ventilator circuit as required including with active humidification
14. Clinician objection.
15. The use or anticipated use of nebulised tobramycin during this clinical episode
16. Any other specific contraindication to anticoagulation including prophylactic anticoagulation not otherwise listed here
17. Relapse in clinical condition in patient that had fully weaned from advanced respiratory support
18. Any systemic anticoagulation other than prophylactic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
D-dimer profile | Up to day 10.
  Effect of nebulised heparin on d-dimer profile, assessed via d-dimer AUC and via a mixed effects model, with data collected on days 1, 3, 5 and 10.
Frequenccy of Severe Adverse Outcomes | Up to day 60
  Safety of nebulised heparin delivered by aerogen solo nebuliser in patients with COVID-19 induced severe respiratory failure, as measured by the incidence of severe adverse events.

SECONDARY OUTCOMES:
Oxygenation Index | Up to day 10
  Determine the impact of nebulised heparin on oxygenation index
Indices of Inflammation | Up to day 10
  Effect of nebulised heparin on indices of inflammation (Interleukin (IL)-1β, IL-6, IL-8, IL-10 and soluble TNF receptor 1 (sTNFR1), C-reactive protein, procalcitonin, Ferritin,) will be assessed (AUC on days 1, 3, 5 and 10)
Ratios of Indices of Inflammation | Up to day 10
  Effect of nebulised heparin on the ratios of IL-1β/IL-10 and IL-6/IL-10 will also be assessed.
Indices of Coagulation | Up to day 10
  Effect of nebulised heparin on other indices of coagulation (Fibrinogen; lactate dehydrogenase) will be assessed (AUC on days 1, 3, 5 and 10).
Quasi-Static Lung Compliance | Up to day 10
  Determine the effect of nebulised heparin on Quasi-Static Lung Compliance (i.e. tidal volume/(Plateau pressure-PEEP) measured on days 1,3,5,10.
Time to separation from advanced respiratory support | Up to day 28
  Time to separation from advanced respiratory support, where non survivors are treated as though not separated from advanced respiratory support.
Number treated with neuromuscular blockers | Up to day 10
  Number treated with neuromuscular blockers instituted after enrolment
Number treated with Prone positioning | Up to day 10
  Number treated with prone positioning instituted after enrolment
Number treated with extra-corporeal membrane oxygenation | Up to day 10
  Number treated with extra-corporeal membrane oxygenation instituted after enrolment
Number requiring Tracheostomy | Up to day 28
  Number tracheotomised
Time to separation from invasive ventilation among survivors | Up to day 28
  Time to separation from invasive ventilation among survivors
Discharge to ward | Up to day 28
  Time to separation from the ICU to day 28, where non-survivors to day 28 are treated as though not separated from invasive care
Discharge to ward in survivors | Up to day 28
  Time to discharge from the ICU to day 28, among survivors
Patient Survival | Up to day 60
  Survival to day 28; Survival to day 60; and Survival to hospital discharge, censored at day 60
Number of patients residing at home or in a community setting at day 60 | Up to day 60
  Number residing at home or in a community setting at day 60
Number of surviving patients residing at home or in a community | Up to day 60
  Number residing at home or in a community setting at day 60, among survivors
Ventilatory ratio | Up to day 10
  Effect of nebulised heparin on ventilatory ratio measured every 6 hours
Number treated with awake prone positioning | Up to day 10
  Number of patients treated with awake prone positioning

CONTACTS AND LOCATIONS:
Overall Officials: John Laffey, Principal Investigator — Professor of Anaesthesia and Intensive Care Medicine, National University of Ireland, Galway, Ireland
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Investigator will consider requests to share anonymised data for the purposes of meta-analysis following discussion with the sponsor.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Investigator will consider release of the above data once the study report has been completed.
Access Criteria: To be confirmed, prior to enrollment of the first patient.

REFERENCES:
- [Derived] Sheehan JR, Calpin P, Kernan M, Kelly C, Casey S, Murphy D, Alvarez-Iglesias A, Giacomini C, Cody C, Curley G, McGeary S, Hanley C, McNicholas B, van Haren F, Laffey JG, Cosgrave D. The CHARTER-Ireland trial: can nebulised heparin reduce acute lung injury in patients with SARS-CoV-2 requiring advanced respiratory support in Ireland: a study protocol and statistical analysis plan for a randomised control trial. Trials. 2022 Sep 14;23(1):774. doi: 10.1186/s13063-022-06518-z. PMID 36104785